CLINICAL TRIAL: NCT01684462
Title: A Phase IIB Placebo Comparative, Double Blinded, Randomized, Multi-center Study to Evaluate the Efficacy and Safety of ALbumin Therapy in Acute Ischemic Stroke Patients in Korea.
Brief Title: The Efficacy and Safety Study of ALbumin Therapy in Acute Ischemic Stroke
Acronym: ALbumin
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul St. Mary's Hospital (Other)
Collaborators: Green Cross Corporation (Industry)
Responsible Party: Principal Investigator, Kwang Soo Lee, Neurology Professor, Seoul St. Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AL_IIT_01
Record Dates: First submitted 2012-08-21; First posted 2012-09-13 (Estimated); Last update posted 2013-12-02 (Estimated); Status verified 2013-11

CONDITIONS: Cerebral Infarction
Keywords: Acute Ischemic Stroke; Albumin
MeSH Terms: conditions — Cerebral Infarction; Ischemic Stroke | interventions — Serum Albumin, Human; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Human Serum Albumin 20 (Experimental): Human Serum Albumin 20% 100cc intravenously infused over 4~8h
  Interventions: Biological: Human Serum Albumin 20
- 0.9 % Normal saline (Placebo Comparator): Treatment with same volume of normal saline
  Interventions: Drug: 0.9 % Normal Saline

INTERVENTIONS:
Biological: Human Serum Albumin 20 — Human Serum Albumin 20% 100cc albumin 1.25g/kg up to 100g (500ml) intravenously infused over 4~8h, commencing within 12 hours of stroke onset
  Other Names: Human Serum Albumin Injection 20% 100ml Greencross
  Arms: Human Serum Albumin 20
Drug: 0.9 % Normal Saline — Infusion of 100 mL of 0.9% Normal Saline ( equivalent volume of Albumin ) over 4~8h, commencing within 12 hours of stroke onset
  Other Names: 0.9 % Normal Saline ChoongWae INJ. 100ml
  Arms: 0.9 % Normal saline

SUMMARY:
In this clinical study, the efficacy and safety of ALbumin is to be evaluated for the patients occurred within 12 hours of acute ischemic stroke.

DETAILED DESCRIPTION:
According to the statistics of the cause of death in 2008 by the Statistics Korea, the stroke was accounted for a large proportion of cause of death among adults, as well as higher mortality, severe sequelae. These stroke in acute phase showed neurological deterioration over 50% of the patients after beginning of treatment and the sequelae resulting in that the nervous tissue was not regenerated is regarded as irreversible changes.

The test group administered 20% albumin based on 1.25g/kg (up to 100g (500ml) over 80kg body weight) to the patients occurred within 12 hours of the onset of symptoms and equal amount of placebo (saline solution (0.9% normal saline)) administered to the control group will be compared to evaluate the efficacy and safety of ALbumin for the patients with acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age less than 75 years old
* Patients who can be administered ALbumin within 12hours of onset of acute ischemic stroke
* 5 ≤ NIHSS score < 15
* Patients who are agreed by guardian or legal representative in case that patients have no ability to join study voluntarily

Exclusion Criteria:

* Medical history of congestive heart failure or patients who are judged congestive heart failure on admission.
* Patients with cardiac edema or pulmonary edema.
* Medical history of myocardial infarction within the past six months.
* Patients who have serious aortic stenosis and mitral valve stenosis.
* Signs or symptoms of acute MI on admission (Serum troponin level ≤0.1 ug/L)
* Those Who had cardiac surgery.
* Onset of cerebral infarction within the past three months.
* Before onset of cerebral infarction, patients who were diagnosed as Historical mRS ≥ 2.
* Patients who received treatment of thrombolysis or who planned for treatment of thrombolysis.
* Acute tachyarrhythmia or bradyarrhythmia with hemodynamic instability on admission.
* Acute or chronic lung disease requiring supplemental O2 therapy on admission
* Severe anemia (Hb < 8.0)
* Severe dehydration (defined as decreased skin turgor, dry oral mucous membrane, tachycardia(>100/min), and oliguria)
* Fever, defined as core body temperature>37.5 ℃
* Serum creatinine > 2.0 mg/dL
* History of allergy to albumin.
* Patients who have side effects of albumin (hyperergia to shock, fever, facial flushing,urticarial, algor, lumbodynia)
* Pregnancy
* Patients who are in life-threatening or stupor coma situation.
* Evidence of intracranial hemorrhage (intracerebral hematoma (ICH), subarachnoid hemorrhage (SAH), epidural hemorrhage, acute or chronic subdural hematoma (SDH)) on admission CT or MRI scan.
* Patients who are not the normal, excesses of circulating blood.
* Haemolytic anemia, anemia due to blood loss.
* Immunodeficiency disease, immunosuppression.
* Blood pressure higher than 180/110 mmHg on admission.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-09; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Average change in NIHSS | at 14±3days
  Comparison of the average change in NIHSS between the control and ALbumin group at screening(-12h~0days) and 14±3days

SECONDARY OUTCOMES:
NIHSS Score | at 14±3days
  Comparison of NIHSS score between the control and ALbumin group at 14±3days
Proportion of patients with improvement by NIHSS | at 14±3days
  Comparison of the proportion of patients with improvement in NIHSS over 4 at 14±3days.
modified Rankin Scale(mRS) favorable outcome | at 3 months
  Comparison of the global functional outcome on modified Rankin Scale(mRS) at screening(-12h~0days) and 3 months.
Volume difference on diffusion MRI | at 4 days±1days
  Comparison of the volume difference of cerebral infraction defined by diffusion MRI at 4±1days
Recurrent new ischemic lesions on diffusion MRI | at 4±1days
  Comparison of the proportion of patients who appear to be recurrent new ischemic lesions defined by diffusion MRI

CONTACTS AND LOCATIONS:
Overall Officials: Kwang Soo Lee, M.D, Ph.D, Principal Investigator — Seoul St. Mary's Hospital
Locations (4):
- South Korea (4):
  - St. Vincent's hospital, Suwon, Gyeonggido
  - Ewha Womans University Mokdong Hospital, Mokdong, Seoul
  - Seoul St. Mary's Hospital, Seocho-Gu, Seoul
  - Yeoudo St. Mary's hospital, Yeongdeungpo-gu, Seoul